CLINICAL TRIAL: NCT01697917
Title: A Pilot Randomized Controlled Trial Examining the Differences of Quality of Life of Patients Undergoing Total Gastrectomy or Proximal Gastrectomy for Adenocarcinoma of Esophagogastric Junction
Brief Title: Impact on Quality of Life in Patients Undergoing Total Gastrectomy or Proximal Gastrectomy for Adenocarcinoma of Esophagogastric Junction
Acronym: GCQOL01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yanong Wang, Director of Department of Abdominal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-44-562
Record Dates: First submitted 2012-09-29; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Adenocarcinoma of Esophagogastric Junction.
Keywords: Adenocarcinoma of Esophagogastric Junction; Total Gastrectomy; Proximal Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total Gastrectomy or Proximal Gastrectomy (Other)
  Interventions: Other: Total Gastrectomy or Proximal Gastrectomy

INTERVENTIONS:
Other: Total Gastrectomy or Proximal Gastrectomy

SUMMARY:
The purpose of this study is to find out more about differences of the quality of life in patients undergoing total gastrectomy or proximal gastrectomy for adenocarcinoma of esophagogastric junction. To find a better reconstruction for patients who received total gastrectomy.

DETAILED DESCRIPTION:
Overall, the incidence of stomach cancer worldwide is declining with geographical variation. However, an increase in the incidence rate of adenocarcinoma of esophagogastric junction, called cardia or AEG has been observed in recent years. AEG may represent a specific histopathological and biologic entity. In the treatment AEG there is argument over whether proximal gastractomy(PG) or total gastractomy (TG) should be done. The quality of life (QOL) of the patients following TG or PG arouses people's attention. The purpose of this study was to evaluate differences of the quality of life in patients undergoing total gastrectomy or proximal gastrectomy for adenocarcinoma of esophagogastric junction.

ELIGIBILITY:
Inclusion Criteria:

* • Pathologically confirmed gastric malignant tumor at FUSCC (biopsy may be performed at other institutions but slides must be confirmed at FUSCC, as is routine care at our institution), and the patients be assessed can achieve R0 radical dissection through total gastrectomy or proximal gastrectomy by three specialists.

  * Patients 20-75 years old
  * Normal organ function, able to tolerate surgery, no clear contraindication for surgery
  * No evidence of metastases of adjacent organs
  * be able to provide follow-up over 2 years
  * No specific treatment for gastric cancer before surgery
  * In line with the Declaration of Helsinki and the requirements of the hospital ethics committee.
  * The subjects were able to understand and comply with the trial protocol, and signed informed consent.

Exclusion Criteria:

* • AEG SiewertⅠtype patients

  * Synchronous or metachronous (less than five years) and patients with other malignancies.
  * Cirrhosis and portal hypertension
  * Associated with blood diseases
  * Serious heart/ lung and kidney dysfunction or with metabolic diseases such as diabetes, hyperthyroidism.
  * Suffering from a serious neurological disease or psychological diseases affecting the life.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in QOL (Quality of Life) | 5years
  From preoperative following gastrectomy, as measured with the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-STO22 questionnaires.

SECONDARY OUTCOMES:
Nutritional status of patients | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China